CLINICAL TRIAL: NCT01515631
Title: Characterization of Pulmonary Artery Stenoses in Alagille Syndrome - a Medical Record
Brief Title: Characterization of Pulmonary Artery Stenoses in Alagille Syndrome - a Medical Record Review
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey A. Feinstein, Principal Investigator, Stanford University
Other Study IDs: AG9031
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Alagille Syndrome
MeSH Terms: conditions — Alagille Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study: Patients with alagille syndrome

SUMMARY:
Patients who have Alagille Syndrome (AGS) also frequently have blockages (or "stenoses") of their pulmonary arteries. Little is known about the degree or variability of these stenoses, or the effect of this disease on the right ventricle (the chamber of the heart which pumps blood to the lungs). This study will first quantify and describe pulmonary artery stenosis in patients with Alagille Syndrome. The study will also assess the effect of these stenoses on the right ventricle. The investigators hope to learn the degree and characteristics of pulmonary artery stenosis in Alagille Syndrome. The investigators also hope to learn the effect of this pulmonary artery stenosis on the right ventricle in patients with Alagille Syndrome. This information is critical in the management of patients with Alagille syndrome, as there is currently no data to guide clinicians on the management of pulmonary artery stenosis. Furthermore, the information from this study may help physicians manage pulmonary artery stenosis in other patients as well.

DETAILED DESCRIPTION:
The investigators hope to learn the degree and characteristics of pulmonary artery stenosis in Alagille Syndrome. We also hope to learn the effect of this pulmonary artery stenosis on the right ventricle in patients with Alagille Syndrome. This information is critical in the management of patients with Alagille syndrome, as there is currently no data to guide clinicians on the management of pulmonary artery stenosis. Furthermore, the information from this study may help physicians manage pulmonary artery stenosis in other patients as well. For the third aim, we hope to learn about the different blood vessel abnormalities in the brain, and which abnormalities are most likely to lead to stroke.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Alagille Syndrome

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Alagille Syndrome. The age range will be from birth through adulthood. There will be no gender or ethnic limitations to study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-04; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Assessment of PA in Alagille Patient | Open

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Feinstein, MD, MPH, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No